CLINICAL TRIAL: NCT04401605
Title: Effects of a Fermented Food-Supplemented on Patients with Ulcerative Colitis
Brief Title: Fermented Food-Supplemented Diet in Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Assistant Professor of Medicine (Gastroenterology and Hepatology), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 55558
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases; Diet Modification; Ulcerative Colitis
Keywords: IBD; Ulcerative Colitis; UC; Diet; Fermented Food
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fermented Food-Supplemented Diet (Experimental): Patients in this arm will supplement their regular diet by an increasing number of daily servings of fermented food over a period of 10 weeks.
  Interventions: Other: Fermented Food-supplemented Diet
- Regular Diet Control Arm (Placebo Comparator): Patients in this arm will continue their regular diet throughout the 10 weeks of study with a maximum of 1 serving of fermented foods per day.
  Interventions: Other: Regular Diet

INTERVENTIONS:
Other: Fermented Food-supplemented Diet — Fermented foods include Kimchi, Sauerkraut, Yoghurt, Kefir and more.
  Arms: Fermented Food-Supplemented Diet
Other: Regular Diet — No change in diet.
  Arms: Regular Diet Control Arm

SUMMARY:
The purpose of this study is to see how a diet that supplements fermented foods effects inflammation and quality of life in patients with mild to moderate Ulcerative Colitis (UC). There is a paucity of research and an enormous need for better understanding of diet and intestinal inflammation. Fermented food have been shown to positively influence inflammatory cytokines and intestinal microbial diversity in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female subjects, ≥18 years of age
* Confirmed diagnosis of UC
* Symptomatic disease defined as partial Mayo Score 2 to 7 (inclusive)
* Elevated fecal calprotectin

Exclusion Criteria:

* Women who are pregnant, nursing or expect to be pregnant
* Intolerance to fermented food
* Individuals with a body mass index (BMI) lower than 18
* Individuals diagnosed with a serious medical condition (unless approved in writing by a physician)
* Individuals who have been severely weakened by a disease or medical procedure
* Individuals with more than mild-moderate cardiovascular disease or life-threatening cancer (as determined by patient's physician) unless approved by a physician
* Individuals with history of severe cardiac disease (particularly uncompensated congestive heart failure NYHA grade 2 or more or LVEF < 40%)
* History of relevant intestinal surgery such as total or hemi-colectomy, proctocolectomy, stoma.

Complications of disease such as extraintestinal manifestations (EIMs) are not automatically considered exclusion criteria. Appropriate medical treatment for UC and/or EIMs will not be withheld.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in the clinical disease activity inflammatory marker fecal calprotectin | Baseline (Data Collection 1) versus Week 10 (Data Collection 2).
  Change in fecal calprotectin

SECONDARY OUTCOMES:
Clinical response as per partial Mayo score. | Baseline (Data Collection 1) versus Week 10 (Data Collection 2).
  Clinical response as per partial Mayo score is defined as a decrease from baseline in the partial Mayo Score of >=2 points and either a rectal bleeding subscore of <=1 or a decrease in the rectal bleeding subscore of >=1 point (assessed at Data Collection 2). The partial Mayo score consists of the subscores for stool frequency, rectal bleeding, and PGA, omitting endoscopy. Each subscore is graded from 0 to 3 (3 being the worst situation and 0 the best) and the partial Mayo score is graded from 0 to 9 (0 being the best, 9 being the worst outcome).
Clinical remission as per partial Mayo score. | Assessed at Week 10 (Data Collection 2).
  Clinical remission as per partial Mayo score is defined as a partial Mayo score < 2 points and no individual subscale score >1 point (assessed at Data Collection 2). The partial Mayo score is graded from 0 to 9 (0 being the best, 9 being the worst outcome).
Symptomatic remission as per Patient Reported Outcome (PRO2) score | Assessed at Week 10 (Data Collection 2).
  Symptomatic remission is defined as as a Mayo stool frequency subscore of 0 or 1 and a Mayo rectal bleeding subscore of 0 (assessed at Data Collection 2). The partial Mayo score is graded from 0 to 9 (0 being the best, 9 being the worst outcome).
Patient global assessment | Assessed at Week 10 (Data Collection 2).
  "Do you believe you are in remission from your UC symptoms?" (Yes/No)
Effect of Fermented Food-Supplemented Diet on patient quality of life | Baseline (Data Collection 1) versus Week 10 (Data Collection 2).
  Change in Short Inflammatory Bowel Disease questionnaire (SIBDQ) score. The SIBDQ is a quality of life score in UC patients. Response to each of the questions is graded from 1 to 7 (1 being the worst situation and 7 the best).
Changes in cytokines/chemokines and immune cell profiles | Baseline (Data Collection 1) versus Week 10 (Data Collection 2).
  Cytokines/chemokines (e.g. TNF-alpha, IL-6, IL-10, IFN-gamma, α4β7, CCR1, and CCR9) and immune cell profiles.
Changes in gut microbiome profiles | Baseline (Data Collection 1) versus Week 10 (Data Collection 2).
  Gut microbiome profiles

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No